CLINICAL TRIAL: NCT01792674
Title: A Randomised Educational Feasibility Trial: 'In Situ Simulation' Versus 'Off Site Simulation' in Obstetric Emergencies and the Effect on Knowledge, Safety-attitudes, Team Performance, Stress, and Motivation
Brief Title: 'In Situ Simulation' Versus 'Off Site Simulation' in Obstetric Emergencies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Principal Investigator, Jette Led Sorensen, MD, Consultant Obstetric Gynecologist, MMEd, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: ob-an-op-simulation-trial
Record Dates: First submitted 2013-01-30; First posted 2013-02-15 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Education; Obstetrics; Simulation; 'In Situ Simulation'
Keywords: Education; Patient simulation; In situ simulation; Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- In situ simulation (Experimental): 'In situ simulation' which is training in the actual patient care unit, in this situation the labour suite and operation theatre
  Interventions: Other: In situ simulation
- Off site simulation (Active Comparator): The control group will receive the same training 'off site simulation', i.e., in training rooms away from the actual patient care unit.
  Interventions: Other: Off site simulation

INTERVENTIONS:
Other: In situ simulation
  Arms: In situ simulation
Other: Off site simulation
  Arms: Off site simulation

SUMMARY:
Care for pregnant is a field where unexpected emergencies occur, however emergencies are rare and hence competences difficult to learn. Therefore, it can be relevant to use simulation-based medical education. Many questions on how simulation can optimise learning remain unanswered. A major question is how simulation settings as 'in situ simulation' (i.e. in the actual patient care unit) versus 'off site simulation' (i.e. in training rooms or simulation center) impact learning.

Objectives: To study the effect of 'in situ simulation' versus 'off site simulation' on learning outcome, safety-attitudes, team performance and clinical performance in the simulated setting plus stress and motivational inducing effect of simulation settings.

Design: Randomised trial. Primary outcome: Written knowledge-test. Exploratory outcomes: Safety Attitudes Questionnaire, team- and clinical performance score, validated stress inventory, salivary cortisol, Intrinsic Motivation Inventory and questionnaire on perceptions of the simulation and organisational changes needed.

Perspective: To provide new knowledge on contextual effects of different simulation settings.

DETAILED DESCRIPTION:
Background: Care for pregnant and delivering women is a field where unexpected emergencies, as for example emergency caesarean sectio, postpartum bleeding or severe preeclampsia, that may potentially harm both mother and baby, occur. Obstetric emergencies are rare and hence by nature difficult to learn in real life. Therefore, it can be relevant with simulation-based medical education, i.e., training with mannequins and scenarios. In non-systematic reviews it is concluded that repetitive medical simulations are associated with improved learner outcomes. However, many questions on how simulation can optimise learning in emergencies remain unanswered; e.g., how different kinds of simulation settings as 'in situ simulation' versus 'off site simulation' impact learning at the individual and the team level.

Objectives: In a randomised trial on authentic obstetric-anaesthesia teams to study the effect of 'in situ simulation' versus 'off site simulation' on participants learning outcome, safety-attitudes, team performance plus motivational and stress inducing effect of different simulation settings and the potential association with learning and performance.

Interventions: The experimental intervention is training in 'in situ simulation' which means training in the actual patient care unit, in this situation the labour suite and operation theatre. The control group will receive the same training 'off site simulation', i.e., in training rooms away from the actual patient care unit. In the two different simulation settings, the same scenarios will be conducted and the participants will comprise of authentic teams of specialised obstetricians or obstetric trainees in their final training year, trainee obstetricians, midwifes, auxiliary nurses, specialised anaesthetists or anaesthesia trainees in their final training year, trainee anaesthetists, anaesthesia nurses, and surgical nurses.

Design and trial size: Single-centre investigator-initiated randomised superiority trial. We have chosen to calculate the required sample size based on experiences about knowledge tests. We assume a standard deviation at 24%, and a difference in the experimental and control means at 17%. With alpha set at 0.05, beta set at 0.80 and intraclass correlation at 0,05 the sample size added up to 93 participants. It is planned to include 100 participants.

Outcomes: Primary outcome: 1) Knowledge by written test as multiple choice questions.

Exploratory outcomes: 1) Safety Attitudes Questionnaire SAQ). 2) Team performance score measured by Team Emergency Assessment Measure (TEAM). 3) Clinical performance in the simulated setting. 4) Salivary cortisol. 5) Validated stress inventory (Stress-Trait Anxiety Inventory (STAI-1) and cognitive appraisal). 6) Intrinsic Motivation Inventory (IMI). 7) Questionnaire to evaluate participants' perceptions of the simulation, the debriefing, and changes needed at the organisational level.

Time schedule: 2 years with start planning 1st of April 2012. Randomisation will start after approval from the Regional Ethics Committee and the Danish Data Protection Agency. The intervention with 'in situ simulation' versus 'on site simulation' described in this protocol will be scheduled spring 2013.

ELIGIBILITY:
Inclusion Criteria:

* Health-care professionals (specialised obstetricians, trainee obstetricians, midwifes, auxiliary nurses, specialised anaesthetists, trainee anaesthetists, anaesthesia nurses, and surgical nurses) employed at the Obstetric or Anaesthesia departments at Rigshospitalet and trainee doctors having part of their training programme at Juliane Marie Centre for children, women and reproduction, Rigshospitalet.
* Participants shall work in the evening-, night- and weekend-shift duties with some of their work in labour ward
* Provide signed informed consent before randomisation

Exclusion Criteria:

* Manager with staff responsibilities. Staff taking part in planning of the intervention.
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Knowledge test by written test as multiple-choice questions (MCQ). | The participants will get a knowledge test at the training day they will participate in. Ten training days will be conducted in a 3 months period
  The intervention will be applied on ten training days. Each training day will include training of one authentic team consisting of ten health care professionals.

SECONDARY OUTCOMES:
Exploratory outcomes: Safety Attitudes Questionnaire (SAQ). | The participants will answer the Safety Attitudes Questionnaire (SAQ) 3-6 weeks before and 3-6 weeks after the training day they will participate in. Ten training days will be conducted in a 3 months period.
  Safety Attitudes Questionnaire (SAQ) is an inventory used in several countries. Safety Attitudes Questionnaire (SAQ) is an exploratory outcomes.
Exploratory outcomes: Team Emergency Assessment Measure (TEAM). | Video's will be recorded at the ten training days (within a 3 months period) and within approximately 4 months after the video's will be assessed by independent observers.
  Team performance score measured by Team Emergency Assessment Measure (TEAM) will be assessed by independent observers by reviewing video recordings of the scenarios. A validated rating scale (Cooper S, 2010) will be used. Team Emergency Assessment Measure (TEAM) is an exploratory outcomes.
Exploratory outcomes: Video assessment: Clinical performance in the simulated setting. | Video's will be recorded at the ten training days (within a 3 months period) and within approximately 4 months after be assessed by independent observers.
  Clinical performance in the simulated setting will be assessed by independent observers by reviewing video recordings of the simulations. The assessment will be based on international and national guidelines of best medical practice. Clinical performance in the simulated setting is an exploratory outcomes.
Exploratory outcome: Salivary cortisol | Participants will have testing for salivary cortisol before and after the two simulated scenarios that will be conducted on the training they will participate in.
  Salivary cortisol is an exploratory outcome
Exploratory outcome: State-Trait Anxiety Inventory (STAI-1). | Participants will respond on State-Trait Anxiety Inventory (STAI-1) before and after the two simulated scenarios that will be conducted on the training day they will participate in.
  State-Trait Anxiety Inventory (STAI-1) is a validated stress inventory. State-Trait Anxiety Inventory (STAI-1) is an exploratory outcome.
Exploratory outcome: Cognitive appraisal (CA). | Participants will respond on cognitive appraisal (CA) before and after the two simulated scenarios that will be conducted on the training day they will participate in on one training day.
  Cognitive appraisal (CA) is applied on 10-point Likert scales to get information of the participants perceived stress of the upcoming event along with their capacity to cope with the stressor. Cognitive appraisal (CA) is an exploratory outcome.
Exploratory outcome: Intrinsic Motivation Inventory (IMI). | The participants will answer on Intrinsic Motivation Inventory (IMI) approximately one week after the training day they will have participated in
  Intrinsic Motivation Inventory (IMI) is a validated inventory.Intrinsic Motivation Inventory (IMI) is an exploratory outcome.
Exploratory outcome: Participant's perceptions of the simulations. | The participants will answer on questionnaires about their perceptions of the simulations approximately one week after the training day they will have participated in.
  Participant's perceptions of the simulations will be obtained on questionnaires including questions on Likert scales and few open questions about personal perceptions of the simulations and whether the simulations inspired to changes in the organisation.

CONTACTS AND LOCATIONS:
Overall Officials: Jette Led Sørensen, MD, MMEd, Principal Investigator — Juliane Marie Centre for Children, Women and Reproduction , Rigshospitalet, Copenhagen University Hospital
Locations (1):
- Rigshospitalet, Juliane Marie Centre for Children, Women and Reproduction, Copenhagen, Denmark

REFERENCES:
- [Derived] Fransen AF, van de Ven J, Banga FR, Mol BWJ, Oei SG. Multi-professional simulation-based team training in obstetric emergencies for improving patient outcomes and trainees' performance. Cochrane Database Syst Rev. 2020 Dec 16;12(12):CD011545. doi: 10.1002/14651858.CD011545.pub2. PMID 33325570
- [Derived] Sorensen JL, van der Vleuten C, Rosthoj S, Ostergaard D, LeBlanc V, Johansen M, Ekelund K, Starkopf L, Lindschou J, Gluud C, Weikop P, Ottesen B. Simulation-based multiprofessional obstetric anaesthesia training conducted in situ versus off-site leads to similar individual and team outcomes: a randomised educational trial. BMJ Open. 2015 Oct 6;5(10):e008344. doi: 10.1136/bmjopen-2015-008344. PMID 26443654
- [Derived] Sorensen JL, Van der Vleuten C, Lindschou J, Gluud C, Ostergaard D, LeBlanc V, Johansen M, Ekelund K, Albrechtsen CK, Pedersen BW, Kjaergaard H, Weikop P, Ottesen B. 'In situ simulation' versus 'off site simulation' in obstetric emergencies and their effect on knowledge, safety attitudes, team performance, stress, and motivation: study protocol for a randomized controlled trial. Trials. 2013 Jul 17;14:220. doi: 10.1186/1745-6215-14-220. PMID 23870501
- See also: Related Info — http://rh.dk/simulation-jmc
- Available data/document: Clinical Study Report — http://ncbi.nlm.nih.gov/pmc/articles/PMC4611309/pdf/bmjopen-2015-008344.pdf — Sørensen JL, van der Vleuten C, Rosthøj S, Østergaard D, LeBlanc V, Johansen M, Ekelund K, Starkopf L, Lindschou J, Gluud C, Weikop P, Ottesen B.Simulation-based multiprofessional obstetric anaesthesia training conducted in situ versus off-site leads to similar individual and team outcomes: a randomised educational trial. BMJ Open 2015;5: e008344
- Available data/document: Qualitative study based on the study population from randomised trial. — http://ncbi.nlm.nih.gov/pmc/articles/PMC4608174/pdf/bmjopen-2015-008345.pdf — Sørensen JL, Navne LE, Martin HM, Ottesen B, Albrectsen CK, Pedersen BW. Clarifying the learning experiences of healthcare professionals with in situ versus off site simulation-based medical education: a qualitative study. BMJ Open 2015;5:e008345